CLINICAL TRIAL: NCT01938534
Title: Prospective Study : Helicobacter Pylori Eradication Therapy in Accordance With Past Antibiotics Use
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Sun Gyo Lim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AJOU-EIRB-152692
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Helicobacter Eradication

ARMS (2):
- Experimental (Experimental): Omeprazole 30mg twice Clarithromycin 500mg twice Amoxicillin 1000mg twice
  for 10 days
  Interventions: Drug: Helicobacter pylori eradication
- Control (Active Comparator): Tetracycline 500mg four times Omeprazole 30mg twice Bismuth 600mg twice Metronidazole 500mg three times for 10 days
  Interventions: Drug: Helicobacter pylori eradication

INTERVENTIONS:
Drug: Helicobacter pylori eradication

SUMMARY:
Prospective study : Helicobacter pylori eradication therapy in accordance with past antibiotics use.

DETAILED DESCRIPTION:
Antibiotics resistant is serious problem in helicobacter pylori eradication. Clarithromycin is very important antibiotics in eradication. But clarithromycin resistance is increased. Major cause of clarithromycin resistance is past consumption of macrolide. Thus the investigators propose eradication of macrolide used group bismuth contained four drugs therapy.

ELIGIBILITY:
Inclusion Criteria:

* Peptic ulcer disease
* Gastric MALT lymphoma
* Early gastric cancer
* Familial history of gastric cancer
* Idiopathic iron deficiency
* Chronic idiopathic thrombocytopenia
* Atrophic gastritis
* Helicobacter infected dyspepsia
* Long term NSAIDs use

Exclusion Criteria:

* Pregnant
* Previous proton pump inhibitor, antibiotics or anticoagulant use within 2 weeks
* Previous stomach surgery
* Severe ill patients (heart failure, hepatic failure, renal failure, hematologic disorder, severe psychologic or neurologic disorder)
* Previous Helicobacter eradication
* Allergy for Helicobacter eradication medicine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, South Korea